CLINICAL TRIAL: NCT04121806
Title: Diet Intervention as a Prebiotic Treatment for Active Ulcerative Colitis
Brief Title: Diet Intervention Treatment for Active Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-0112-A; 3U01DK062423-18S1 (NIH)
Record Dates: First submitted 2019-09-30; First posted 2019-10-10 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ulcerative colitis patients with mild to moderate activity (Experimental): Participants will be followed for 14 days on their traditional diet followed by an 8 week intervention with the specially designed and provided treatment diet.
  Interventions: Other: UC intervention diet

INTERVENTIONS:
Other: UC intervention diet — The treatment diet has been designed based on the literature with the goal of influencing the biodiversity and density of the microbiome. All food through the duration of the 8 week dietary intervention period of the study will be provided to the treatment arm study participants.

SUMMARY:
The purpose of this study is to determine if a sustainable non-elemental diet can be used as a probiotic tool to alter the dysbiotic microbiome found in individuals with ulcerative colitis and thereby decrease disease activity.

DETAILED DESCRIPTION:
The etiology of inflammatory bowel disease (IBD), including ulcerative colitis (UC), is complex and poorly understood, but the current hypothesis is that IBD arises from an aberrant immune response to commensal bacteria in a genetically susceptible host, and is triggered by environmental factors. Environmental factors such as the microbiome and diet, play a significant role in the risk of IBD. Diet has been identified as one of the main drivers of the microbiome composition and the microbiome and diet can work in tandem to affect host physiology.

In spite of patient interest in diet and numerous diet studies, currently there is no diet that is clinically validated or universally agreed upon for adult IBD patients. We also lack rigorous studies to show how the microbiome is influenced by diet and affects patient outcomes.

We propose to use a sustainable non-elemental diet aimed at altering the microbiome in patients with mild to moderately active UC to alter their disease activity.

ELIGIBILITY:
Inclusion Criteria:

* • Females and Males between the ages of 18 - 75 years of age at the time of enrolment

  * Must have established diagnosis of UC by standard endoscopic, radiographic, or histological criteria
  * Must have active UC defined by having a Mayo score equal to or greater than 2 within two months prior to enrollment
  * Must have had > 10cm involvement at some point in their disease history
  * FCP>250 or active endo within 6 months
  * If a smoker, must not change smoking habits (frequency) during the course of the study
  * If receiving medical therapy, no baseline therapy change within 4 weeks of study initiation and no change during the course of the study

Exclusion Criteria:

* • Uncontrolled inflammation which will likely require surgery or escalation of therapy within 4 weeks of enrollment

  * Pregnant or lactating females
  * Allergy or intolerance to key or a great number food components of the study diet
  * Current NSAID use
  * Diagnosed with PSC
  * Using topical therapies or suppositories
  * Antibiotic use within 4 weeks of the study enrollment or during the study
  * Confirmed C. difficile infection within 3 months of recruitment;
  * Diagnosis of primary PSC;
  * Currently using topical therapies or suppositories
  * History of dysplasia or colorectal neoplasia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in microbiome composition | 10 weeks
  measured by 16S rDNA sequencing and comparing pretreatment diet and the treatment diet within an individual
Change in microbiome function | 10 weeks
  measured by shotgun sequencing and comparing difference in enriched functional pathways between pretreatment diet and the treatment diet within an individual

SECONDARY OUTCOMES:
Decrease in endoscopic disease activity | 10 weeks
  measured by a decrease in Mayo score between pretreatment diet and the treatment diet within an individual
Decrease in clinical disease activity | 10 weeks
  measured by a decrease in serum C-reactive protein (CRP) levels between pretreatment diet and the treatment diet within an individual

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Study results or individual subject results such as investigational tests will not be shared with the research participants or others unless deemed medically necessary. Result of this research and management of intellectual property will adherence to the NIH Grant Policy on Sharing of Unique Research Resources including the Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources issued March 5, 2003.
  Publication of data during the project and/or at the end of the project shall be consistent with normal scientific practices. Research data which documents, supports, and validates research findings will be made available after the main findings from the final research data set have been accepted for publication.